CLINICAL TRIAL: NCT05706493
Title: Association Between Severity of Periodontitis and the Level of Anti-citrullinated Protein Antibodies (ACPAs) in Rheumatoid Arthritis Patients
Brief Title: Association Between Periodontitis and the Level of Anti-citrullinated Protein Antibodies in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Other Study IDs: PER 3312007
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Diseases; Rheumatoid Arthritis
Keywords: periodontitis; rheumatoid arthritis; anti citrullinated protein antibodies; peptidyl arginine deminase enzyme; gingival crevicular fluid (GCF)
MeSH Terms: conditions — Periodontal Diseases; Arthritis, Rheumatoid; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-surgical periodontal treatment: assessment of different periodontal parameters and gingival crevicular fluid sampling will be done then non surgical periodontal treatment will be performed then after 3 months re assessment of the periodontal parameters and gingival crevicular fluid sampling will be done

SUMMARY:
the relationship between rheumatoid arthritis and periodontal disease is crucial and has been explained via a complex interplay of genetic, environmental, and hormonal factors that influence the host immune tolerance leading to both disease characteristics. The aim of this study is to clinically investigate the correlation between the levels of anti-citrullinated protein antibodies (ACPAs) in gingival crevicular fluid before and after non-surgical periodontal treatment and the severity of periodontal disease and rheumatoid arthritis in rheumatoid arthritis (RA) patients

DETAILED DESCRIPTION:
the relationship between rheumatoid arthritis and periodontal disease is crucial and has been explained via a complex interplay of genetic, environmental, and hormonal factors that influence the host immune tolerance leading to both disease characteristics.

The aim of this study is to clinically investigate the correlation between the levels of anti-citrullinated protein antibodies (ACPAs) in gingival crevicular fluid before and after non-surgical periodontal treatment and the severity of periodontal disease and rheumatoid arthritis in rheumatoid arthritis (RA) patients Materials and Methods: a total of 40 participants suffering from periodontitis and rheumatoid arthritis will be referred from the Badr Hospital (Faculty of Medicine, Helwan University) to Misr international university's dental clinic complex. Gingival crevicular fluid (GCF) samples will be collected from the patients before performing periodontal therapy (baseline). Assessment of ACPAs will be quantified using enzyme-linked immunoassay (ELISA) as the primary outcome at baseline and after 3 months. Assessment of 2ry outcomes includes clinical periodontal and RA parameters at baseline and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid patients fulfilling the ACR criteria for the classification of RA

  * 18 years
* Both genders
* Presence of at least 8 teeth

Exclusion Criteria:

* Smoking
* Diabetes Mellitus
* Pregnant females
* Patients who had undergone periodontal treatment within last 3 months
* Antibiotic therapy during last 3 months
* Other autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid patients
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the level of anti-citrullinated protein antibodies (ACPAs) | at baseline and 3 months
  assessment of the level of anti-citrullinated protein antibodies (ACPAs) in gingival crevicular fluid

SECONDARY OUTCOMES:
Change in Clinical attachment Loss | at baseline and 3 months
  measuring the distance from the cemento enamel junction to the base of the pocket in mm
Change in Probing depth | at baseline and 3 months
  measuring the distance from the gingival margin to the base of the pocket in mm
Change in Plaque index (PI) | at baseline and 3 months
  it is a score (0,1,2 and 3) where: 0 = No plaque in the gingival area. 1 = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface. 2 = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye. 3 = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Hafez, Lecturer, Principal Investigator — Lecturer, faculty of oral and dental medicine misr international university; Yahia Hassan, Lecturer, Principal Investigator — Lecturer, faculty of oral and dental medicine misr international university; Shahinaz Al ashiry, asso.Prof, Study Director — Associate Professor, faculty of oral and dental medicine misr international universit
Locations (1):
- Faculty of oral and dental medicine, Misr international university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No